CLINICAL TRIAL: NCT01331135
Title: Sirolimus in Combination With Metronomic Therapy in Children With Recurrent and Refractory Solid Tumors: A Phase I Study
Brief Title: Aflac ST0901 CHOANOME - Sirolimus in Solid Tumors
Acronym: Aflac ST0901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Muna Qayed, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047016; Aflac ST0901 CHOANOME (Other: Other)
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Ewing's Sarcoma; Osteosarcoma; Astrocytoma; Atypical Teratoid/Rhabdoid Tumor; Ependymoma; Germ Cell Tumor; Glioma; Medulloblastoma; Rhabdoid Tumor; Retinoblastoma; Clear Cell Sarcoma; Renal Cell Carcinoma; Wilms Tumor; Hepatoblastoma; Neuroblastoma; Rhabdomyosarcoma
Keywords: pediatrics; sirolimus; relapse
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma; Astrocytoma; Rhabdoid Tumor; Ependymoma; Neoplasms, Germ Cell and Embryonal; Glioma; Medulloblastoma; Retinoblastoma; Sarcoma, Clear Cell; Carcinoma, Renal Cell; Wilms Tumor; Hepatoblastoma; Neuroblastoma; Rhabdomyosarcoma; Recurrence | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sirolimus treatment (Experimental): Dose escalation of sirolimus with starting dose at 1 mg/m2 and increasing to a possible 3 mg/m2.
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — daily administration of sirolimus in oral form starting at a dose of 1 mg/m2 and increasing to a possible 3 mg/m2.
  Other Names: rapamune; cypher; renacept

SUMMARY:
The best treatment for recurrent cancers or those that do not respond to therapies is not known. Typically, patients with these cancers receive a combination of cancer drugs (chemotherapy), surgery, or radiation therapy. These treatments can prolong their life but may not offer a long-term cure.

This study proposes using a drug called Sirolimus in combination with common chemotherapy drugs to treat patients with recurrent and refractory solid tumors. Sirolimus has been found to inhibit cell growth and to have anti-tumor activity in pediatric solid tumors in previous studies and, therefore, has the potential to increase the effectiveness of the chemotherapy drugs when given together.

This study wil investigate the highest dose of Sirolimus that can be given orally with other oral chemotherapy drugs. Cohorts of 2 subjects will be started at the minimum dose. The dose will be increased in the next 2 subjects as long as there were no major reactions in the previous groups. This study will also seek to learn more about the side effects of sirolimus when used in this combination and what effects the drug has on the white cells and the immune system. Successful use of this drug will impact the cancer population greatly by providing an increased chance of survival to those with resistant or recurrent cancers.

DETAILED DESCRIPTION:
Sirolimus, is a potent immunosuppressive drug that is approved for use in prevention against allograft rejection following solid organ transplant. It has anti-tumor effects mainly by blocking signals which drive cells from G1 to S phase during cell cycle through inhibition of mTOR, thus inhibiting cell growth. Sirolimus, as well as other mTOR inhibitors, has shown anti-tumor activity in pediatric solid tumor xenografts. Children with relapsed and/or refractory solid tumors are in need of novel therapeutic approaches. One option for these patients is the use of prolonged exposure to low dose antiangiogenic chemotherapy, with agents such as etoposide and cyclophosphamide. In this phase I trial the feasibility and optimal dosing for daily sirolimus, in combination with daily celecoxib, and low dose etoposide alternating with cyclophosphamide, will be determined in children with relapsed and refractory solid tumors. p70S6 kinase inhibition will be used as a surrogate for mTOR inhibition. The potential immunosuppressive effect of sirolimus administered on this schedule will be assessed by serial lymphocyte subsets and assessment of memory T cell number.

ELIGIBILITY:
Inclusion Criteria:

* must be <=30 years of age at time of study enrollment
* histologic verification of malignancy at original diagnosis or relapsis except in patients with intrinsic brain stem tumors, optic pathway gliomas or patients wtih pineal tumors and evaluations of serum or CSF alpha-fetoprotein or beta-HCG
* measurable or evaluable disease
* disease state must be one for which there is no known curative therapy
* Performance level >=50%
* Patients must have fully recovered from acute toxic effects of all prior chemotherapy, immunotherapy or radiotherapy
* no evidence of acute graft vs. host disease and >=3 months since transplant
* organ function as defined in eligibility section of protocol

Exclusion Criteria:

* patients cannot be pregnant or breast-feeding
* patients must agree to use of an effective contraceptive method
* no growth factors that support platelet or white cell number or function for at least 7 days prior to enrollment
* patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the prior 7 days are not eligible
* patients receiving any other investigational drugs
* patients receiving any other anti-cancer drugs
* patients who have an uncontrolled infection

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years after treatment starts
  estimate the maximum tolerated dose (MTD) and recommended Phase II dose of sirolimus administered orally once daily for 42 days in combination with metronomic chemotherapy in children with recurrent or refractory solid tumors.

SECONDARY OUTCOMES:
define and describe toxicities of sirolimus | 2 years post treatment
  To define and describe the toxicities of sirolimus administered in combination with metronomic chemotherapy administered according to this schedule.
anti-tumor activity of sirolimus | 2 years post treatment
  To assess the antitumor activity of sirolimus administered in combination with metronomic chemotherapy to children with recurrent and refractory solid tumors within the confines of a Phase I study.
evaluate correlation of p70S6 kinase activity | 2 years post treatment
  To evaluate the correlation of p70S6 kinase activity inhibition with tumor response.
evaluate risk of infection | 2 years post treatment
  To evaluate the effect of this combination therapy on lymphocyte subsets and memory T-cells, and to correlate that with risk of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Qayed, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Result] Qayed M, Cash T, Tighiouart M, MacDonald TJ, Goldsmith KC, Tanos R, Kean L, Watkins B, Suessmuth Y, Wetmore C, Katzenstein HM. A phase I study of sirolimus in combination with metronomic therapy (CHOAnome) in children with recurrent or refractory solid and brain tumors. Pediatr Blood Cancer. 2020 Apr;67(4):e28134. doi: 10.1002/pbc.28134. Epub 2019 Dec 25. PMID 31876107
- See also: Clinical trials website for Children's Healthcare of Atlanta — http://www.choa.org/Childrens-Hospital-Services/Cancer-and-Blood-Disorders/Research/Clinical-Trials/Find-a-Clinical-Trial